CLINICAL TRIAL: NCT02329418
Title: Impact of a Written Document on Post Traumatic Stress Disorder (PTSD) Diagnosed in Family Members After Withholding and Withdrawing Life-sustaining Therapies in the Intensive Care Unit
Brief Title: Written Document to Assist Family During Decision of Withholding and Withdrawing Life-sustaining Therapies in the Intensive Care Unit
Acronym: LATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-A00758-39
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written document (Experimental): Accompanying relatives with a written document when discussing withholding and withdrawing life-sustaining therapies . All other procedures are standard.
  Interventions: Other: Explaining withholding and withdrawing life-sustaining therapies along with a written document
- Standard (Active Comparator): Discussing withholding and withdrawing life-sustaining therapies following standard procedure without written document
  Interventions: Other: Explaining withholding and withdrawing life-sustaining therapies following standard procedure

INTERVENTIONS:
Other: Explaining withholding and withdrawing life-sustaining therapies along with a written document — The document describes the law and the role of family members and medical team in the decision.
  Arms: Written document
Other: Explaining withholding and withdrawing life-sustaining therapies following standard procedure
  Arms: Standard

SUMMARY:
Relatives of patients in situation of withholding and withdrawing life-sustaining therapies often show post traumatic stress disorder (PTSD) (60%)[1]. This number is even greater when family members are active in this decision (81%) or when communication is not optimal between medical team and family members.

There are several ways to assist families of patients in intensive care units [2], amongst them the use of a written document to explain the environment, therapies and possible outcomes.

Here the investigators want to test the impact of a written document in the context of end-of-life conference in intensive care units. Specifically, this research addresses wether such written support could decrease 3-months post-traumatic stress disorder, anxiety and depression exhibited by the closest family member or the patient representative.

ELIGIBILITY:
The study will enroll patient representant (family member or close friends designed by the family or pre-admission legal representant).

Inclusion Criteria:

* Medical team anticipates a decision to withhold and withdraw life-sustaining therapies to intensive care unit (ICU) discharge
* verbal consent to participate
* Able to communicate in French

Exclusion Criteria:

* representant of a patient < 18 years old
* representant of a patient whose stay in ICU lasted less than 48 hours
* representant of a patient without social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Rate of PTSD | 3 months
  PTSD is assessed with Impact Event Scale (IES) on the family representative

SECONDARY OUTCOMES:
Rate of depression | 3 months
  Depression is assessed with Hospital Anxiety and Depression scale (HADS) on the family representative
Rate of anxiety | 3 months
  Anxiety is assessed with Hospital Anxiety and Depression scale (HADS) on the family representative
Mean level of HADS (anxiety and depression subscales) | 3 months
Mean level of IES | 3 months
Length of the processus from decision to withhold and withdraw life-sustaining therapies to intensive care unit (ICU) discharge | An average of 6 days
Respectfulness of the law regarding withholding and withdrawing life-sustaining therapies | An average of 6 days
Rate of decision to withhold and withdraw life-sustaining therapies in different intensive care units from the hospital | ICU discharge (an average of 3 weeks)
Medical Doctor satisfaction with the processus | ICU discharge (an average of 3 weeks)
Description of the processus | ICU discharge (an average of 3 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Critical Care Depratment, Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Schmidt M, Azoulay E. Having a loved one in the ICU: the forgotten family. Curr Opin Crit Care. 2012 Oct;18(5):540-7. doi: 10.1097/MCC.0b013e328357f141. PMID 22914431
- [Derived] Robin S, Labarriere C, Sechaud G, Dessertaine G, Bosson JL, Payen JF. Information Pamphlet Given to Relatives During the End-of-Life Decision in the ICU: An Assessor-Blinded, Randomized Controlled Trial. Chest. 2021 Jun;159(6):2301-2308. doi: 10.1016/j.chest.2021.01.072. Epub 2021 Feb 5. PMID 33549600